CLINICAL TRIAL: NCT05841134
Title: Multicenter, Single-arm, Open-label Phase II Clinical Study of Tislelizumab Combined With Chemotherapy (CAPOX) in the Perioperative Treatment of MSI-H/dMMR Stage II or III Colorectal Cancer
Brief Title: Tislelizumab Combined With Chemotherapy (CAPOX) in the Perioperative Treatment of MSI-H/dMMR Stage II or III Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Head of the oncology ward, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-CAPOX-MSI-H-CRC-
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: MSI-H Colorectal Cancer; Tislelizumab; Oxaliplatin; Capecitabine
MeSH Terms: interventions — tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with CAPOX (Experimental): Successfully screened subjects will receive 4 cycles of neoadjuvant therapy with tislelizumab combined with chemotherapy (CAPOX) before surgery； undergo radical surgery 4-6 weeks after the end of the last medication; tislelizumab will be given after surgery Monoclonal antibody ± chemotherapy adjuvant therapy (the investigator judges whether to add chemotherapy based on the patient's comprehensive condition), until disease progression or unacceptable toxicity, the longest treatment is 12 months.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Neoadjuvant treatment options:
  Tislelizumab 200mg, intravenous infusion, D1, Q3W, a total of 4 cycles; Oxaliplatin 130mg/m2, intravenous infusion, D1, Q3W, 4 cycles in total; Capecitabine 1000mg/m2, orally twice in the morning and evening, D1-14, Q3W, 4 cycles in total;
  Adjuvant treatment options:
  Tislelizumab 200mg, intravenous infusion, Q3W;
  ± Chemotherapy method (researcher judges whether to add chemotherapy according to the comprehensive condition of the patient); Until disease progression or unacceptable toxicity, the maximum treatment time is 12 months.
  Other Names: Capecitabine; Oxaliplatin

SUMMARY:
This study is a multi-center, single-arm, open-label phase II clinical trial, aiming to observe and evaluate the perioperative treatment of tislelizumab combined with chemotherapy (CAPOX) in stage II or III colorectal cancer with MSI-H/dMMR Patient efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG: 0~1;
2. Patients with colon or rectal adenocarcinoma confirmed by histology or cytology;
3. The tissue specimens are confirmed as MSI-H by PCR or NGS. If the patients are dMMR by immunohistochemistry, they need to be confirmed as MSI-H by PCR (2021 Expert Consensus on Immunotherapy for Patients with Colorectal Cancer);
4. Patients with clinical stage II or III (cT3-T4 N0 M0 or Tany N+M0, clinically positive lymph nodes are defined as any lymph node ≥ 1.0 cm);
5. Expected survival period ≥ 12 weeks;
6. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with follow-up visits.

Exclusion Criteria:

1. Have received anti-tumor therapy;
2. Have received PD-(L)1 or CTLA-4 treatment;
3. The patient has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis , hyperthyroidism; patients with vitiligo; asthma that has been completely remitted in childhood and does not require any intervention in adulthood can be included; patients with asthma requiring medical intervention with bronchodilators cannot be included);
4. Patients are using immunosuppressants or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other equivalent hormones), and continue to use within 2 weeks before enrollment;
5. Patients with any severe and/or uncontrolled diseases
6. Urine routine prompts urine protein ≥ ++, and confirmed 24-hour urine protein quantity > 1.0g;
7. Pregnant or lactating women;
8. Patients with other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
9. Those who have a history of psychotropic drug abuse and cannot quit or patients with mental disorders;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) | Up to 24 months
  After receiving tislelizumab combined with CAPOX neoadjuvant, the rate of pathological complete remission (after neoadjuvant therapy, for those who insist on organ preservation, combined with imaging and endoscopic examination to achieve cCR, and the biopsy result of the microscope is pathological Complete remission can be judged as pCR)

SECONDARY OUTCOMES:
R0 resection rates | Up to 24 months
  The proportion of patients achieved a complete resection with negative margin.
Overall survival (OS) | Up to 36 months
  Defined as the time from randomization to death from any cause.
Event-free survival (EFS) | Up to 36 months
  Event-free survival is the time from the beginning of enrollment to the occurrence of any event, including death, disease progression, change to chemotherapy, change to chemotherapy, addition of other treatments, and occurrence of fatal or intolerable side effects
Incidence of adverse events during the treatment and follow-up (safety) | until 100 days after last patient last study drug treatment
  Adverse events will be assessed during treatment and follow-up.